CLINICAL TRIAL: NCT05075252
Title: REsiDENT1 (Re-assessment of Appendicitis Evaluation During Laparoscopic Appendectomy: Do we End a Non-standardized Treatment Approach and Habit?): Peritoneal Irrigation During Laparoscopic Appendectomy-Does the Grade of Contamination Matter? A Prospective Multicenter Resident-based Evaluation of a New Classification System
Brief Title: Re-assessment of Appendicitis Evaluation During Laparoscopic Appendectomy, Peritoneal Irrigation During Laparoscopic Appendectomy Does the Grade of Contamination Matter?
Acronym: RESIDENT1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S_26_05_21_5158
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Appendicitis; Appendectomy
Keywords: laparoscopy; appendicitis; appendectomy; lavage; suction; abscess
MeSH Terms: conditions — Appendicitis; Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- R1: patients affected by acute appendicitis undergoing totally laparoscopic appendectomy
  Interventions: Procedure: laparoscopic lavage

INTERVENTIONS:
Procedure: laparoscopic lavage — This study aims to investigate the impact of laparoscopic lavage on the incidence of postoperative abscesses stratifying patients on the grade of appendicitis and peritoneal contamination.

SUMMARY:
Type: prospective observational multicenter trial. Population of interest: adult patients undergoing laparoscopic appendectomy for acute appendicitis.

Hypothesis : laparoscopic lavage during laparoscopic appendectomy is a practice that should be used in selected patients according to the intraperitoneal grade of contamination and grade of appendicitis. Nonregulated use of laparoscopic lavage cannot be considered superior to suction only considering recent evidence. Few RCT available addressing this issue are available, but any with a high methodological quality.

Aim: The aim of this study is to investigate the impact of laparoscopic lavage during laparoscopic appendectomy on the postoperative incidence of intrabdominal abscesses, stratifying patients in different clusters according to a defined classification considering the intraperitoneal contamination and grade of appendicitis.

DETAILED DESCRIPTION:
Introduction: Laparoscopic appendectomy has progressively gained acceptance as the standard of care for acute appendicitis. Focusing on the incidence of postoperative intra-abdominal abscess after a laparoscopic appendectomy, discordant data have been reported ranging from 1.5 to 20%. Besides, evidence advocating advantages from peritoneal irrigation over suction only are lacking. Most studies are burdened by a high level of heterogeneity regarding the severity of the appendicitis and modalities of peritoneal irrigation. One of the main drawbacks is the lack of an accepted classification for different degrees of appendicitis and peritoneal contamination. The aim of the study is to introduce a classification to clarify the relationship between grade of appendicitis, contamination, and postoperative incidence of IAA considering the surgeon's attitude toward irrigation or suction alone. Preoperative, intra-operative, and postoperative predictive factors for infectious complication will also be assessed. This study is meant to be the first Italian multicenter resident-based observational study.

Hypothesis: The driving hypothesis of the investigators study is that there should exist a relationship between different intra-operative treatment protocols (irrigation vs suction alone) and postoperative incidence of IAA. Furthermore, considering various grades of appendicitis and peritoneal contamination, the use of irrigation vs suction alone could lead to different rates of postoperative IAA.

Aim: The aim of this study is to introduce and evaluate a classification for acute appendicitis taking into account the peritoneal contamination to delineate the relationship between grade of appendicitis and postoperative incidence of IAA considering the surgeon's attitude toward irrigation or suction alone.

Primary endpoint:

Relationship among each severity grade of acute appendicitis and postoperative incidence of intra-abdominal abscesses

Secondary endpoint:

Impact of intraperitoneal irrigation or suction alone on the incidence of IAA for each severity grade

Methods:

See the dedicated section for eligibility criterion. Participants will fill an online form reporting all clinical and intra-operative data of each patient who will undergo a laparoscopic appendectomy. All personal information of patients will be removed according to data anonymization.

Data will be reported in accordance with Strengthening the Reporting of Observational studies in Epidemiology guidelines (STROBE) for observational studies [22].

Residents from each involved center will be responsible for data collection. All forms will be collected in an electronic database by the coordinating residents who will check for data completeness. All residents taking part in the study will be asked to enter eventual missing data.

The incidence of IAA after laparoscopic appendectomy reported in the literature ranges from 1.5 to 20% [4, 5, 9,10,11]. Such a wide interval is not negligible when calculating the sample size (n) of the study cohort. Furthermore, some important basic considerations need to be taken into account: appendicitis is the most common acute surgical disease so the baseline population is large and cannot be exactly estimated; the incidence of intra-abdominal abscesses has never been systematically investigated in regard to the severity of appendicitis and contamination. All patients included in the study will be classified into different clusters considering the grade of appendicitis and contamination, lavage vs suction alone, and postoperative incidence of IAA.

Considering all these aspects, sample size for power calculation can be reasonably estimated given a 95% confidence interval with a z-score of 1.96, a 50% standard deviation, and a 0.03 margin of error. This formula does not include the incidence rate of IAA for the aforementioned reasons.

The estimated sample size would be around at least 1067 patients. Data will be collected in a computerized spreadsheet (Microsoft Excel 2016; Microsoft Corporation, Redmond; WA) and analyzed with statistical software (IBM Corp. Released 2017. IBM SPSS Statistics for Windows, version 25.0. Armonk, NY).

χ2 test will be assessed to compare categorical variables, and univariate logistic regression will be performed to provide hazard ratios for individual variables, identifying possible predictors of postoperative complication (IAA above all). All significant (p < 0.05) variables at univariate analysis will be included in a multivariate regression model in order to detect independent risk factors for the outcome and to estimate odds ratio and 95% confidence intervals.

A scoring system will be built according to the results of statistical analysis. The weight of each variable will be addressed based on odds ratio values. To evaluate the accuracy of the score, discrimination and calibration of the model will be explored. The former will be assessed by receiver operating characteristic (ROC) curve analysis, whereas the latter will be investigated with the Hosmer-Lemeshow goodness-of-fit test. Based on the results of the ROC curve analysis, we will proceed to identify different severity grades of acute appendicitis each one related to a specific risk of developing delayed IAA. χ2 test will be assessed to compare categorical variables, and univariate logistic regression will be performed to provide hazard ratios for individual variables, identifying possible predictors of postoperative complication (IAA above all). All significant (p < 0.05) variables at univariate analysis will be included in a multivariate regression model in order to detect independent risk factors for the outcome and to estimate odds ratio and 95% confidence intervals.

Discussion The observational nature of this study is mandatory to examine and analyze surgeon attitude toward peritoneal contamination related to appendicitis during laparoscopic appendectomy. The optimal study design to address the core matter would be a well-structured RCT to assess the real effect of lavage plus suction versus suction alone on postoperative IAA. There is a lack of methodological strictness in the existent randomized trials due to heterogeneous determination of appendicitis severity and peritoneal contamination.

We feel indispensable to start from identifying different grades of appendicitis, related contamination, and their relationship with postoperative abscesses, considering surgeons' attitude. The core step is to classify each patient and create a score to pick out classes of peri-appendiceal contamination related to different incidence rate of postoperative IAA.

The General Surgery residency program at the University of Milan is based on a large clinical network in which residents are distributed in different hospitals. It is a 5-year program. One hundred thirty residents are involved. The clinical network includes 59 surgical units in 27 hospitals.

This system structure allows great exposure to different surgical scenarios, inside and outside the operating room. The program requires, per year, a minimum of procedures in which the resident has to be involved. From the first to the fifth year, the difficulty of the procedure is increased. To the best of the investigators' knowledge, this is one of the most efficient residency programs in Italy because great attention is dedicated to surgical skills improvement. On the other hand, this program may underestimate the scientific needs and educational growth of residents. This study is resident driven as an incitement to a defined organization for the scientific growth of the University of Milan residents.

During the project start-up phase of this study, an official group of residents of the General Surgery program at the University of Milan has been created. The main aim of this group of young doctors is to try to guarantee to each resident, who is interested, the minimal scientific knowledge and ability to critically understand, ideate, and project a scientific study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 69 years old
* Surgical laparoscopic approach for AA
* Intra-operative and histological diagnosis of AA

Exclusion Criteria:

* Patients < 18 years old or > 69 years old
* Previous appendectomy
* Previous appendicitis treated conservatively
* Open approach for surgery or intra-operative conversion
* Co-existence of other intra-abdominal infections (IAI)
* Patients with immunodeficiency
* Patients treated with steroid, immunosuppressant, or CHT within previous 6 months

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing laparoscopic appendectomy for acute appendicitis
Sampling Method: Probability Sample
Enrollment: 1067 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Intrabdominal Abscess | 90 days after surgery
  Surgical site infections are divided into three categories: superficial incisional SSI,deep incisional SSI and organ/space surgical site infection.O/S SSI must meet the following criteria;date of event within 30 days after surgical procedure,involvement of any part of the body deeper than the fascial/muscle layers that are opened or manipulated during the operative procedure.At least one of the following:purulent drainage from a drain that is placed into the organ/space (eg;closed suction drainage system,open drain,T-tube drain,CT-guided drainage).Organism(s) identified from fluid or tissue in the organ/space by a culture- or non-culture-based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment.An abscess or other evidence of infection involving the organ/space that is detected on the gross anatomical or histopathologic exam,or imaging test evidence suggestive of infection

SECONDARY OUTCOMES:
Postoperative complication | 90 days
  Any postoperative complication according to Clavien Dindo classification > 2a

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Cioffi SPB, Altomare M, Spota A, Granieri S, Cimbanassi S, Chiara O. REsiDENT 1 (Re-assessment of Appendicitis Evaluation during laparoscopic appendectomy: Do we End a Non-standardized Treatment approach and habit?): peritoneal irrigation during laparoscopic appendectomy-does the grade of contamination matter? A prospective multicenter resident-based evaluation of a new classification system. World J Emerg Surg. 2019 May 30;14:25. doi: 10.1186/s13017-019-0243-4. eCollection 2019. PMID 31164914
- [Derived] Cioffi SPB, Granieri S, Scaravilli L, Molteni M, Altomare M, Spota A, Virdis F, Bini R, Renzi F, Reitano E, Ragozzino R, Gupta S, Chiara O, Cimbanassi S; Resident-1 Research Group. Surgeons' attitudes during laparoscopic appendectomy: do subjective intraoperative assessments affect the choice of peritoneal irrigation? A spin-off analysis from the REsiDENT-1 multicentre prospective observational trial. Surg Endosc. 2023 Jan;37(1):729-740. doi: 10.1007/s00464-022-09674-0. Epub 2022 Oct 28. PMID 36307601